CLINICAL TRIAL: NCT00564187
Title: Prospective, Multicentric, Randomized, Open, Comparative Phase IV Study Evaluating the Efficacy and Safety of the Dosage Adjustment of Aprovel® (Irbesartan) in Hypertensive Outpatients in Current Clinical Practice
Brief Title: Evaluation of Efficacy and Safety of the Dosage Adjustment of Aprovel® (Irbesartan) in Hypertensive Outpatients in Current Clinical Practice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_8484
Record Dates: First submitted 2007-11-20; First posted 2007-11-27 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Until 6 weeks: 150mg/day, then a dosage adjustment according to the blood pressure(normalized: DBP<90mmHg, responding non normalized:DBP≥90mmHg and a decrease of DBP≥10mmHg, non responding: decrease of DBP<10mmHg and DBP≥90mmHg) for the period between 6 and 12 weeks:
  • 150mg/day for normalized patients and patients responding non normalized randomized in the group A
  Interventions: Drug: Irbesartan
- 2 (Active Comparator): • Or 300 mg/day for non responding patients and responding patients non normalized randomized in the group B
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: Irbesartan — Irbesartan: 150mg tablets
  Dosage: Until 6 weeks: 150mg/day, then a dosage adjustment according to the blood pressure(normalized: DBP<90mmHg, responding non normalized:DBP≥90mmHg and a decrease of DBP≥10mmHg, non responding: decrease of DBP<10mmHg and DBP≥90mmHg) for the period between 6 and 12 weeks:
  • 150mg/day for normalized patients and patients responding non normalized randomized in the group A
  Arms: 1
Drug: Irbesartan — Irbesartan: 150mg tablets
  Until 6 weeks: 150mg/day, then a dosage adjustment according to the blood pressure(normalized: DBP<90mmHg, responding non normalized:DBP≥90mmHg and a decrease of DBP≥10mmHg, non responding: decrease of DBP<10mmHg and DBP≥90mmHg) for the period between 6 and 12 weeks:
  • Or 300 mg/day for non responding patients and responding patients non normalized randomized in the group B
  Arms: 2

SUMMARY:
Primary:

* To evaluate the efficacy of two regimens of irbesartan in patients responding but not normalized at 6 weeks of treatment (schema N°1: maintenance 150 mg/day, schema n°2: 300 mg/day for 6 more weeks)

Secondary:

* To evaluate the percentage of patients with DBP < 90 mmHg at 6 and 12 weeks
* To evaluate the percentage of patients with SBP < 140 mmHg at 6 and 12 weeks
* To evaluate rate of adverse events during the study

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate hypertension (90mmHg<DBP<110mmHg and 140mmHg<SBP<180mmHg)
* Or new diagnosed hypertension (after 2 visits within 1 month), never treated before and responding to required conditions for a treatment with irbesartan, after an adapted but insufficient diet
* Or a patient having already been treated with a non-satisfying antihypertensive treatment stopped since at least 2 weeks before the inclusion
* A minimum exam labs as required by WHO-ISH within the month before the inclusion

Exclusion Criteria:

* Severe Arterial Hypertension (PAS > than or = to 180 mm Hg or PAD > than or = to 110 mmHg)
* Isolated Systolic Hypertension
* Secondary Hypertension
* Bilateral renal arterial stenosis or renal arterial stenosis
* Non surgically sterilised woman or non post-menopausal woman
* Confirmed sodium depletion
* Irbesartan hypersensitivity

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2003-02; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To Evaluate the efficacy of two regimens of irbesartan in patients responding but not normalized (schema N°1: maintenance 150mg/day, schema n°2: 300mg/day for 6 more weeks) | at 6 weeks of treatment

SECONDARY OUTCOMES:
• To evaluate the percentage of patients with DBP<90 mmHg | at 6 and 12 weeks
• To evaluate rate of adverse events | during the study duration
• To evaluate the percentage of patients with SBP<140 mmHg | at 6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chokri Jeribi, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Mégrine, Tunisia